CLINICAL TRIAL: NCT02620878
Title: Use of Artificial Pancreas in Pediatric Patients. Feasibility , Safety and Efficacy Study of an Automatic Control of Blood Glucose 24/24 at a Diabetes Camp
Brief Title: Artificial Pancreas in Pediatric Patients (PEDarPAN)
Acronym: PEDarPAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Daniela Bruttomesso, medical doctor, University of Padova
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3486/AO/15
Record Dates: First submitted 2015-11-18; First posted 2015-12-03 (Estimated); Results first posted 2019-07-12 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-04

CONDITIONS: Type 1 Diabetes
Keywords: Artificial pancreas; SAP therapy; children; adolescents; type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Pancreas, Artificial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AP (Experimental): Experimental arm: A closed-loop control system (artificial pancreas) will be used during night and day for 72 hours (3 days) with the aim of automate insulin infusion by an insulin pump to control glucose level. AP is composed of a CGM device (Dexcom G4), an insulin pump (Accu Chek Spirit combo, Roche), and a model predictive control algorithm that is embedded in a smartphone and wirelessly linked to the CGM device and insulin pump. A remote monitoring will be ensured all the time the AP will be active and study team will be present in the camp.
  Patients will be randomly assigned to receive either 3 days of automated closed-loop insulin delivery (intervention) followed by 3 days of sensor -augmented pump therapy (control), or the inverted sequence
  Interventions: Device: artificial pancreas
- SAP (Active Comparator): Active Comparator: Sensor Augmented Pump (SAP teraphy : CGM + insulin pump) will be used for 72 hours during day and night (3 days).
  Patients will be randomly assigned to receive either 3 days of SAP (Control) followed by 3 days of automated closed-loop insulin delivery (intervention), or the inverted sequence
  Interventions: Other: sensor augmented pump

INTERVENTIONS:
Device: artificial pancreas — Patients will be randomly assigned to receive either 3 days of automated closed-loop insulin delivery (intervention) followed by 3 days of sensor -augmented pump therapy (control), or the inverted sequence.
  Arms: AP
Other: sensor augmented pump — During this control period (comparator arm) the patients will use sensor augmented pump. This period will be compared to the same period of artificial pancreas
  Arms: SAP

SUMMARY:
The purpose of this study is to determine safety, feasibility and efficacy (with respect to sensor- augmented pump therapy) of an Artificial Pancreas (AP) prototype in day and night closed-loop control in children and adolescents with type 1 diabetes.

DETAILED DESCRIPTION:
The AP prototype is based on a Modular Model Predictive Control algorithm (MMPC) implemented on the Diabetes Assistant (DiAs) wearable platform.

The study will be divided in two parts: the first part will serve as a 3 days pilot study and will be conducted in a hotel/residence near the hospital.

The investigators will recruit 6/8 children (5-12 years) and/or 6/8 adolescents (12-18 years), with type 1 diabetes who have experience with insulin pump. DiAs will be used 72 continuous hours of day and night.

If part 1 will be successfully, after about 2-3 months, the study will move to the second part (the main part), that will consist in cross-over randomized study that will be conducted in a camp setting. The participants will be randomly assigned to the treatment arm (Artificial Pancreas) or to the control arm (sensor-augmented insulin pump). Then the same patient will be assigned to the other arm. Each treatment will be applied 3 consecutive days. During the first period (days 1-3) patients will do the same activites and will have the same diet as in the second period (day s 5-7).

The investigators will recruit 30/40 children (5-12 years) and/or 30/40 adolescents (12-18 years), affected by type 1 diabetes who have experience with insulin pump therapy.

The study has the permission of the Ethics Committee reference and the permission for "clinical investigation with devices not CE marked" by the Health Ministry.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of type 1 diabetes · The diagnosis of type 1 diabetes is based on the investigator's judgment

   · C peptide levels and antibody determinations are not required
2. Daily insulin therapy for ≥ 12 months
3. Insulin pump therapy for ≥ 3 months
4. Age 6-18 years
5. A1C<10
6. Avoidance of acetaminophen-containing medications (i.e. Tachipirina, tachidol, tachiflu) while wearing the continuous glucose monitor.
7. Willingness to wear a continuous glucose sensor
8. Female subjects who are sexually active must be on acceptable method of contraception (e.g. oral contraceptive pill, diaphragm, IUD).

Exclusion Criteria:

1. Diabetic ketoacidosis in the past month
2. Hypoglycemic seizure or loss of consciousness in the past 3 months
3. History of seizure disorder (except for hypoglycemic seizure)
4. A1C>10
5. History of any heart disease including coronary artery disease, heart failure, or arrhythmias
6. Cystic fibrosis
7. Current use of oral glucocorticoids, beta-blockers or other medications, which in the judgment of the investigator would be a contraindication to participation in the study.
8. History of ongoing renal disease (other than microalbuminuria).
9. Subjects requiring intermediate or long-acting insulin (such as NPH, Detemir , Glargine or Degludec).
10. Subjects requiring other anti-diabetic medications other than insulin (oral or injectable).
11. Pregnancy - verbal denial of pregnancy obtained with telephone informed consent, pregnancy test performed at camp before study devices are assigned.
12. Sexually active females who do not practice acceptable contraceptive methods to prevent pregnancy.
13. Presence of a febrile illness within 24 hours of admission or acetaminophen use while wearing the CGM. The subject may be rescheduled for Research House/hotel admission if these criteria are not met. The camp study subject will not participate in the trial if these conditions are met.
14. Medical or psychiatric condition that in the judgment of the investigator might interfere with the completion of the protocol such as:

    * Inpatient psychiatric treatment in the past 6 months
    * Uncontrolled adrenal insufficiency
    * Alcohol abuse

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2015-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Bruttomesso, MD, Principal Investigator — University of Padova, Italy
Locations (1):
- University of Padova, Padua, Italy

REFERENCES:
- [Derived] Del Favero S, Boscari F, Messori M, Rabbone I, Bonfanti R, Sabbion A, Iafusco D, Schiaffini R, Visentin R, Calore R, Moncada YL, Galasso S, Galderisi A, Vallone V, Di Palma F, Losiouk E, Lanzola G, Tinti D, Rigamonti A, Marigliano M, Zanfardino A, Rapini N, Avogaro A, Chernavvsky D, Magni L, Cobelli C, Bruttomesso D. Randomized Summer Camp Crossover Trial in 5- to 9-Year-Old Children: Outpatient Wearable Artificial Pancreas Is Feasible and Safe. Diabetes Care. 2016 Jul;39(7):1180-5. doi: 10.2337/dc15-2815. Epub 2016 May 10. PMID 27208335

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Loop Than Closed Loop: Patients used for 3 days subcutaneous delivery of insulin according to usual pump regimen (open loop), than artificial pancreas for 3 days
- Closed Loop Than Open Loop: Patients used for 3 days artificial pancreas, than subcutaneous delivery of insulin according to usual pump regimen (open loop) for 3 days
Period: Overall Study
Arm/Group | Open Loop Than Closed Loop | Closed Loop Than Open Loop
Started (participants in "CLOSED LOOP First" are also being counted in the "OPEN LOOP Second") | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Experimental arm: A closed-loop control system (artificial pancreas) will be used during night and day for 72 hours (3 days) with the aim of automate insulin infusion by an insulin pump to control glucose level. AP is composed of a CGM device (Dexcom G4), an insulin pump (Accu Chek Spirit combo, Roche), and a model predictive control algorithm that is embedded in a smartphone and wirelessly linked to the CGM device and insulin pump. A remote monitoring will be ensured all the time the AP will be active and study team will be present in the camp.
  artificial pancreas: Patients will be randomly assigned to receive either 3 days of automated closed-loop insulin delivery (intervention) followed by 3 days of sensor -augmented pump therapy (control), or the inverted sequence.
Arm/Group | All Study Participants
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.6 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 32
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Italy | 32

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time Spent With Blood Glucose < 3.9 mmol/L (or 70 mg/dl)
Description: percentage of time spent in hypoglicemia (< 70 mg/dl or 3.9 mmol/L) both during day and night.
  All analyses will include a comparison of the results in Artificial Pancreas and SAP period
Time Frame: 3 days
Measure: Mean (Inter-Quartile Range); unit: percentage
Groups:
- CLOSED LOOP: Experimental arm: A closed-loop control system (artificial pancreas) will be used during night and day for 72 hours (3 days) with the aim of automate insulin infusion by an insulin pump to control glucose level. AP is composed of a CGM device (Dexcom G4), an insulin pump (Accu Chek Spirit combo, Roche), and a model predictive control algorithm that is embedded in a smartphone and wirelessly linked to the CGM device and insulin pump. A remote monitoring will be ensured all the time the AP will be active and study team will be present in the camp.
  artificial pancreas: Patients will be randomly assigned to receive either 3 days of automated closed-loop insulin delivery (intervention) followed by 3 days of sensor -augmented pump therapy (control), or the inverted sequence.
- OPEN LOOP: Active Comparator: SAP teraphy (CGM + insulin pump) will be used for 72 hours during day and night (3 days).
  sensor augmented pump: During this control period (comparator arm) the patients will use sensor augmented pump. This period will be compared to the same period of artificial pancreas
Arm/Group | CLOSED LOOP | OPEN LOOP
Number analyzed (Participants) | 30 | 30
percentage | 2 [1.2 to 4.5] | 6.7 [2.3 to 11.5]

2. Primary Outcome: Percentage of Time Spent in Target Range (70-180 mg/dl or 3.9-10.0 mmol/L)
Description: percentage of time spent in target range (70-180 mg/dl or 3.9-10.0 mmol/L) both during day and night.
  All analyses will include a comparison of the results in Artificial pancraes and SAP period
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | CLOSED LOOP | OPEN LOOP
Number analyzed (Participants) | 30 | 30
percentage | 56.8 (13.5) | 63.1 (11)

3. Secondary Outcome: Percentage of Time Artificial Pancreas is Active
Description: percentage of time that the system worked without any technical problem
Time Frame: 3 days
Measure: Mean (Inter-Quartile Range); unit: percentage of time
Arm/Group | CLOSED LOOP
Number analyzed (Participants) | 30
percentage of time | 97 [93.5 to 98.4]

ADVERSE EVENTS:
Arm/Group | CLOSED LOOP | OPEN LOOP
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No